CLINICAL TRIAL: NCT03644303
Title: TRAP - Targeted Radiotherapy in Androgen-suppressed Prostate Cancer Patients.
Brief Title: Targeted Radiotherapy in Androgen-suppressed Prostate Cancer Patients.
Acronym: TRAP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Collaborators: Prostate Cancer UK (Other); University College, London (Other); The Christie NHS Foundation Trust (Other); The Leeds Teaching Hospitals NHS Trust (Other); Velindre NHS Trust (Other Government); University Hospital Birmingham NHS Foundation Trust (Other); Newcastle-upon-Tyne Hospitals NHS Trust (Other); Belfast Health and Social Care Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCR 4781
Record Dates: First submitted 2018-08-15; First posted 2018-08-23 (Actual); Last update posted 2019-11-14 (Actual); Status verified 2019-11

CONDITIONS: Prostate Cancer; Metastasis; Toxicity Due to Radiotherapy; Circulating Tumour DNA
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasm Metastasis | interventions — Radiosurgery; Androgen Antagonists; enzalutamide; abiraterone

STUDY DESIGN:
Intervention Model Description: Single arm, prospective interventional cohort study
Masking Description: Interpretation of the two paired WB DW MRI scans (baseline and 6 months) will be conducted by one assessor will be blinded to the identity of the baseline scan to ensure minimisation of any potential bias.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SBRT + ADT (Experimental): Enzalutamide OR Abiraterone at licensed doses in combination with stereotactic radiotherapy: 30 Gray in 5 fractions
  Interventions: Radiation: SBRT + ADT

INTERVENTIONS:
Radiation: SBRT + ADT — Short course SBRT to 1 or 2 oligo-progressing metastases in addition to continued abiraterone or enzalutamide
  Other Names: Enzalutamide or Abiraterone plus stereotactic radiotherapy

SUMMARY:
This multi-center, phase II trial will be conducted in men with castration resistant prostate cancer. The aim of the TRAP trial is to test whether a new precise radiotherapy technique called stereotactic body radiotherapy (SBRT) can slow down the growth of metastatic prostate cancer. If SBRT is effective it will represent a new treatment option in these patients, providing more prolonged control without having to resort to chemotherapy and its potentially unpleasant side effects.

In this trial, the investigators will identify men who, despite being on next generation androgen deprivation treatment (Abiraterone or Enzalutamide) have developed one or two new sites of worsening (growing) disease but the rest of their cancer is still responding to hormonal therapy. If it is the case that SBRT can successfully treat the cancer which is resistant to current treatment then the investigators hope they will be able to better control the spread of cancer in these patients for longer.

The investigators also hope that they will be able to use the tell-tale products (gene markers) that are released into the bloodstream in these patients, or identify characteristics on novel imaging such as magnetic resonance imaging (MRI) to help identify patients in the future who will benefit the most.

DETAILED DESCRIPTION:
For many men with metastatic prostate cancer, the cancer develops resistance to successive systemic therapies and eventually all treatment options are exhausted and the patient succumbs to their disease. It is therefore vital to find ways of evading prostate cancer resistance. Stereotactic body radiotherapy (SBRT) has the advantage that it destroys cancerous tissue irrespective of the underlying genetic deficit within the progressing metastasis. If the resistant clones are localized to 1-2 metastases and can be destroyed or ablated, the patient can continue to receive the benefit of their systemic (androgen deprivation) treatment (Abiraterone or Enzalutamide) which may continue to control the remainder of their disease for many months, possibly even years.

SBRT is a recognised technique for the elimination of isolated metastases in other tumour sites achieving local control of metastasis in 80-90% of cases. This is achieved with very few side effects. In the TRAP trial, the investigators wish to establish whether it is beneficial to target 1 or 2 metastatic sites with SBRT or whether patients will develop polymetastatic progression. Patients enrolled on the trial will receive 30 Gy in 5 fractions on alternate days over 10 days. They will continue their androgen deprivation treatment throughout and following SBRT. Side effects will be closely monitored throughout and patients will be seen at the end of radiotherapy and then 4 weeks after treatment. Thereafter patients will undergo trial follow up three monthly which will includes Prostate Specific Antigen (PSA) monitoring.

In addition to the above procedures, the investigators will use a combination of whole body (WB) diffusion weighted (DW) magnetic resonance imaging (WB DW MRI) and circulating tumour (ct) deoxyribonucleic acid (DNA), 'ct DNA' biomarker analysis with the aim of identifying those patients which benefit most from the combination of SBRT and androgen deprivation treatment. WB DW MRI is a novel MRI technique which shows improved sensitivity compared to standard MRI. The marker ctDNA enables the investigators to explore genomic characterisation and variation of metastases and compare findings with previously explored genome mutations in prostate cancer patients.

ELIGIBILITY:
Inclusion Criteria:

1. Be willing and able to provide written informed consent for the trial and be ≥18 years of age on day of signing informed consent.
2. Have metastatic Castration Resistant Prostate Cancer (CRPC) based on biochemical or pathological diagnosis and be on Enzalutamide or Abiraterone.
3. Have had a minimum of 6 months on Enzalutamide or Abiraterone with evidence of response (PSA, radiological or symptomatic)
4. Have 1 - 2 metastatic lesions progressing on imaging (CT, bone scan, MRI or other local imaging) or a clinical or imaging diagnosis of progression of a non-irradiated primary site with the remainder of their metastases currently controlled by Enzalutamide or Abiraterone.
5. Have had no previous radical radiation to the index area (defined as unable to deliver SBRT doses in this protocol without taking normal tissues beyond tolerance).
6. Have a Performance Status (PS) assessed using the Eastern Co-operative Oncology Group (ECOG) criteria of 0 - 1.
7. Have an oligoprogressing site, including those that have developed on treatment, in bone, lymph node, prostate or lung but not in liver, brain, adrenal or other sites.
8. Patients may be symptomatic in the oligoprogressing area. However, there is no urgent need to start radiotherapy.

Exclusion Criteria:

1. A clinical need exists to switch therapy immediately (e.g. suspicion of rapid clinical progression, urgent need for palliative radiotherapy).
2. Evidence of previous invasive cancer in the last 5 years, with the exception of non-melanoma skin cancer (non-invasive malignancies such as non-muscle invasive bladder cancer are not excluded).
3. There is a contra-indication to radiotherapy (e.g. inflammatory bowel disease).
4. There is a contra-indication to MRI where required for radiotherapy (e.g. cardiac pacemaker, internal defibrillator, shrapnel injury or claustrophobia).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 84 (Estimated)
Dates: Start 2018-08-13 (Actual); Primary Completion 2020-10-01 (Estimated); Study Completion 2021-10-01 (Estimated)

PRIMARY OUTCOMES:
Median Progression-Free Survival (PFS) | Outcome to be assessed at 6 months from end of SBRT
  Median progression free survival following SBRT to oligo-progressing metastatic sites assessed using the RECIST (v 1.1) criteria on imaging such as computed Tomography (CT),bone scan, magnetic Resonance Imaging (MRI) or Positron Emission Tomography (PET) scan

SECONDARY OUTCOMES:
Local control rate following SBRT | Outcome to be assessed at 6 months and 1 year from end of SBRT
  Overall control defined as stable disease or partial response of irradiated metastases assessed using the RECIST (v 1.1) criteria on imaging such as computed Tomography (CT), magnetic Resonance Imaging (MRI) or Positron Emission Tomography (PET) scan or control on bone scan
Incidence and severity of treatment induced symptoms | From the start of SBRT up to 24 months following delivery of SBRT
  Incidence of acute and late side-effects resulting from SBRT assessed using the Common Terminology Criteria for Adverse Events (CTCAE) and the Radiotherapy and Oncology Group Terminology Criteria for Adverse Events (CTCAE) and the RTOG (Radiotherapy Oncology Group) scoring criteria
Health Related Quality of Life | Change from start of radiotherapy to each time-point including 3 and 6 months after end of SBRT
  Patient Reported Quality of Life assessed using the Euroqual (EQ) EQ-5D-5L questionnaire
Time to administration of next line of therapy | From the end of SBRT up to 24 months following delivery of SBRT
  Survival and median survival prior to alternative therapy administration
Association between selected WB DW MRI characteristics at baseline and prognosis after SBRT | Outcome to be assessed at 6 months and 1 year from end of SBRT
  Correlation or regression analysis of characteristics (e.g. number of metastases)

OTHER OUTCOMES:
Exploration of novel bio-markers to assess response to SBRT treatment | Assessment of Progression Free Survival at 6 months and 1 year
  Levels of circulating tumor Deoxyribonucleic Acid (ctDNA)

CONTACTS AND LOCATIONS:
Overall Officials: Alison Tree, FRCR, Principal Investigator — Royal Marsden NHS Foundation Trust
Locations (7):
- United Kingdom (7):
  - The Christie NHS Foundation Trust, Manchester, Manchester Greater
  - Belfast Health & Social care Trust, Belfast, Northern Ireland
  - The Royal Marsden NHS Foundation Trust, Sutton, Surrey
  - The Newcastle Upon Tyne Hospitals NHS Foundation Trust, Newcastle upon Tyne, Tyne and Wear
  - Velindre Cancer Centre, Cardiff, Wales
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham, West Midlands
  - Leeds Teaching Hospitals NHS Trust, Leeds, West Yorkshire

IPD SHARING:
Plan to Share IPD: Yes
Human tissue (blood) in surplus will be made available for other ethically approved research provided patients have given their informed consent
Time Frame: Not anticipated to be before 6 months have elapsed following recruitment of the last patient.
Access Criteria: On provision of written request

REFERENCES:
- [Derived] Lee J, Koom WS, Byun HK, Yang G, Kim MS, Park EJ, Ahn JB, Beom SH, Kim HS, Shin SJ, Kim K, Chang JS. Metastasis-Directed Radiotherapy for Oligoprogressive or Oligopersistent Metastatic Colorectal Cancer. Clin Colorectal Cancer. 2022 Jun;21(2):e78-e86. doi: 10.1016/j.clcc.2021.10.009. Epub 2021 Nov 18. PMID 34903471